CLINICAL TRIAL: NCT05295446
Title: Functional GI Disease Registry
Acronym: FGIDR
Status: Enrolling by invitation | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2015P002637
Record Dates: First submitted 2022-03-01; First posted 2022-03-25 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to establish a prospective observational cohort of individuals with functional GI disorders (functional constipation, irritable bowel syndrome, chronic nausea, functional diarrhea, and functional dyspepsia, as well as a subset of these individuals starting neuromodulation for their functional GI disorder) and collect clinical information and specimens. This information will be used in order to establish a patient registry with detailed clinical data and a specimen repository for future research as well as to specifically identify environmental, genetic, physiological, and psycho-social factors associated with functional GI disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Rome IV criteria for a functional GI disorder

Exclusion Criteria:

* Acute illness
* Known bleeding disorder
* Awaiting transplantation
* Known diagnosis of Inflammatory Bowel Disease
* Use of antibiotics in last 2 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with a functional GI disorder
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-02-11 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Single Nucleotide Polymorphism (SNP) genotyping | Baseline visit
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Whole genome analysis | Baseline visit
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Proteomics | Baseline visit
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Microbiome analysis | Baseline visit
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Microbiome analysis | 3 months after enrollment
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Microbiome analysis | 6 months after enrollment
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Microbiome analysis | 1 year after enrollment
  In this study, we anticipate identifying differential functional genomic profiles (metagenomes) and metabolites (metabolomes) between patients with different functional GI disorders, with detailed species-specific reconstruction of microbial metabolic pathways, their complement of gene orthologs, taxonomic distributions, and abundance profiles.
Diet and Lifestyle Questionnaire | Baseline visit
  This questionnaire evaluates patients' diet, lifestyle, and symptoms relating to their functional GI disorder.
Diet and Lifestyle Questionnaire | 3 months after enrollment
  This questionnaire evaluates patients' diet, lifestyle, and symptoms relating to their functional GI disorder.
Diet and Lifestyle Questionnaire | 6 months after enrollment
  This questionnaire evaluates patients' diet, lifestyle, and symptoms relating to their functional GI disorder.
Diet and Lifestyle Questionnaire | 1 year after enrollment
  This questionnaire evaluates patients' diet, lifestyle, and symptoms relating to their functional GI disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Staller, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States